CLINICAL TRIAL: NCT02521298
Title: Lateral Elbow Tendinopathy: A Randomized Controlled Trial Examining The Treatment Effect Of Strength Training Combined With Cortico-Steroid Injection, Dry-Needling Or Placebo
Brief Title: Treatment of Lateral Elbow Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Simon Doessing, M.D., PhD, M.D., PhD, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-15002993
Record Dates: First submitted 2015-07-09; First posted 2015-08-13 (Estimated); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Epicondylitis, Lateral Humeral
MeSH Terms: conditions — Tennis Elbow | interventions — Resistance Training; Dry Needling

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Strength Training + Placebo (Active Comparator): Strength Training: 2 weeks after the inclusion, the patients are instructed in heavy slow resistance exercise by a physiotherapist. Exercise is continued 3 times/week for the following 12 weeks, with supervised follow-up at week 4, 8 and 12. Exercise consists of wrist extension, flexion and supination/pronation. Starting at 3 x 15 repetition maximum, gradually increasing in weight to 3 x 6 repetition maximum from week 8.
  Placebo: Ultrasound-guided subcutaneous injection of 2 ml isotonic saline over the proximal part of the common extensor tendon origin using a 0,8 mm needle. No-touch technique is used, and the patient is blinded with regards to the content of the syringe and the ultrasound-image.
  Interventions: Other: Strength Training; Procedure: Placebo
- Strength Training + Cortico-Steroid Inj. (Experimental): Strength Training: 2 weeks after the inclusion, the patients are instructed in heavy slow resistance exercise by a physiotherapist. Exercise is continued 3 times/week for the following 12 weeks, with supervised follow-up at week 4, 8 and 12. Exercise consists of wrist extension, flexion and supination/pronation. Starting at 3 x 15 repetition maximum, gradually increasing in weight to 3 x 6 repetition maximum from week 8.
  Cortico-Steroid Injection: Ultrasound-guided injection of 1 ml depomedrol 40 mg/ml + 1 ml lidocaine 10 mg/ml deep to the proximal part of the common extensor tendon origin using a 0,8 mm needle. No-touch technique is used, and the patient is blinded with regards to the content of the syringe and the ultrasound-image.
  Interventions: Other: Strength Training; Drug: Cortico-Steroid Injection. Depomedrol 40mg/1ml.
- Strength Training + Dry Needling (Experimental): Strength Training: 2 weeks after the inclusion, the patients are instructed in heavy slow resistance exercise by a physiotherapist. Exercise is continued 3 times/week for the following 12 weeks, with supervised follow-up at week 4, 8 and 12. Exercise consists of wrist extension, flexion and supination/pronation. Starting at 3 x 15 repetition maximum, gradually increasing in weight to 3 x 6 repetition maximum from week 8.
  Dry Needling: Ultrasound-guided penetration of the proximal part of the common extensor tendon origin is repeated 10 times using a 0,8 mm needle, followed by subcutaneous injection of 2 ml isotonic saline superficial to the tendon. No-touch technique is used, and the patient is blinded with regards to the content of the syringe and the ultrasound-image.
  Interventions: Other: Strength Training; Procedure: Dry Needling

INTERVENTIONS:
Other: Strength Training
Procedure: Placebo
  Arms: Strength Training + Placebo
Drug: Cortico-Steroid Injection. Depomedrol 40mg/1ml.
  Arms: Strength Training + Cortico-Steroid Inj.
Procedure: Dry Needling
  Arms: Strength Training + Dry Needling

SUMMARY:
This study investigates the treatment effect on lateral elbow tendinopathy of strength training in combination with cortico-steroid injection, dry-needling or placebo in a double-blinded randomized controlled trial.

DETAILED DESCRIPTION:
The prevalence of lateral elbow tendinopathy is prevalence of 1-3%, with a peak incidence between 35-50 years of age (Green et al., 2002). The main symptoms are pain over the lateral humeral epicondyle upon palpation and pain full resisted dorsiflexion of the wrist. Ultrasonographic changes include hyper-/hypo-echoic areas and increased doppler signal in the most proximal part of the common extensor tendon. The condition is often self-limiting, however full recovery often takes months to years and recurrence is common. Several different treatment modalities are used in order to increase tendon healing and decrease time to recovery. Deep transverse friction massage showed no significant effect on pain, grip strength or function relative to other physiotherapy modalities (Brosseau et al., 2002). Anti-inflammatory treatment with NSAID's or corticosteroids is typically effective in the short term, however on a longer term there is a poorer outcome than with other treatment strategies including exercise (Coombes et al., 2010). Surgery does not seem to have any beneficial effect (Buchbinder et al., 2011), and there are no conclusive data regarding the use of orthotic devises for the treatment of lateral elbow tendinopathy (Struijs et al., 2002). Eccentric exercise of the extensor muscles has been shown to reduced pain, increase muscle strength, and decrease tendon thickness and time to return to sport (Croisier et al., 2007).

Loading of human tendon leads to increased tendon collagen synthesis, and interestingly, tendon tissue sampling (biopsies), which causes a minor trauma to the tendon has been shown to increase the level of growth factors locally and stimulate tendon collagen synthesis (Magnusson et al., 2010).

It is hypothesized that both minimal tissue damage and anti-inflammatory treatment could increase tendon healing and decrease time to recovery, when combined with mechanical loading.

ELIGIBILITY:
Inclusion Criteria:

1. Pain around the lateral part of the elbow joint for more than 4 weeks.
2. Pain on palpation of the proximal part of the common extensor tendon.
3. Pain reproduced with resisted dorsiflexion of the wrist.
4. Dash score > 30.
5. Ultrasonographic appearance consistent with lateral elbow tendinopathy (irregular appearance of the tendon, hypo-/hyper-echoic changes, pathological doppler signal, increased tendon thickness).

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) > 2 (mild systemic disease).
* Patients with symptoms consistent with differential diagnoses such as:

  * referred pain,
  * radiohumeral synovitis and bursitis,
  * posterior interosseous nerve entrapment (radial tunnel syndrome),
  * osteoarthritis of the elbow, and
  * prior injections or acupuncture around the elbow joint within the last 6 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-10; Primary Completion 2020-04-05 (Actual); Study Completion 2020-04-05 (Actual)

PRIMARY OUTCOMES:
Change in disability questionnaire: DASH-score. Area under the DASH-score versus time curve (AUC). | Baseline, week 17, 30, and 56.

SECONDARY OUTCOMES:
Change in muscle strength measurements. Area under the strength measurements versus time curve (AUC) | Baseline, week 17, 30, and 56.
  Including isometric wrist extension force and isometric grip strength.
Change in ultrasonographic appearance of tendon pathology associated with tendinopathy. | Baseline, week 30, and 56.
  Week 0-2, 30 and 56. Including: 1) Irregular appearance of the tendon, 2) Hypo-/hyper-echoic changes, 3) Pathological doppler signal, 4) Tendon thickness.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kjaer, M.D., PhD., Study Director — Bispebjerg Hospital, University of Copenhagen
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark

REFERENCES:
- [Background] Green S, Buchbinder R, Barnsley L, Hall S, White M, Smidt N, Assendelft W. Acupuncture for lateral elbow pain. Cochrane Database Syst Rev. 2002;2002(1):CD003527. doi: 10.1002/14651858.CD003527. PMID 11869671
- [Background] Brosseau L, Casimiro L, Milne S, Robinson V, Shea B, Tugwell P, Wells G. Deep transverse friction massage for treating tendinitis. Cochrane Database Syst Rev. 2002;(4):CD003528. doi: 10.1002/14651858.CD003528. PMID 12519601
- [Background] Coombes BK, Bisset L, Vicenzino B. Efficacy and safety of corticosteroid injections and other injections for management of tendinopathy: a systematic review of randomised controlled trials. Lancet. 2010 Nov 20;376(9754):1751-67. doi: 10.1016/S0140-6736(10)61160-9. Epub 2010 Oct 21. PMID 20970844
- [Background] Croisier JL, Foidart-Dessalle M, Tinant F, Crielaard JM, Forthomme B. An isokinetic eccentric programme for the management of chronic lateral epicondylar tendinopathy. Br J Sports Med. 2007 Apr;41(4):269-75. doi: 10.1136/bjsm.2006.033324. Epub 2007 Jan 15. PMID 17224433
- [Background] Magnusson SP, Langberg H, Kjaer M. The pathogenesis of tendinopathy: balancing the response to loading. Nat Rev Rheumatol. 2010 May;6(5):262-8. doi: 10.1038/nrrheum.2010.43. Epub 2010 Mar 23. PMID 20308995
- [Background] Struijs PA, Smidt N, Arola H, Dijk vC, Buchbinder R, Assendelft WJ. Orthotic devices for the treatment of tennis elbow. Cochrane Database Syst Rev. 2002;(1):CD001821. doi: 10.1002/14651858.CD001821. PMID 11869609
- [Derived] Couppe C, Dossing S, Bulow PM, Siersma VD, Zilmer CK, Bang CW, Hoffner R, Kracht M, Hogg P, Edstrom G, Kjaer M, Magnusson SP. Effects of Heavy Slow Resistance Training Combined With Corticosteroid Injections or Tendon Needling in Patients With Lateral Elbow Tendinopathy: A 3-Arm Randomized Double-Blinded Placebo-Controlled Study. Am J Sports Med. 2022 Aug;50(10):2787-2796. doi: 10.1177/03635465221110214. Epub 2022 Jul 22. PMID 35867777